CLINICAL TRIAL: NCT06255002
Title: Concordance Between the Measurement of Whole Blood Fibrinogen by the qLabs®FIB Analyzer and Its Measurement by Conventional Method (Clauss Fibrinogen) in the Context of Severe Postpartum Haemorrhage: a Prospective Multicenter Non-interventional Study
Brief Title: Concordance Between the Measurement of Whole Blood Fibrinogen by the qLabs®FIB Analyzer and Its Measurement by Conventional Method (Clauss Fibrinogen) in the Context of Severe Postpartum Haemorrhage
Acronym: FIB-HPPS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231640
Record Dates: First submitted 2023-12-05; First posted 2024-02-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Postpartum Hemorrhage
Keywords: Severe postpartum haemorrhage; Fibrinogen concentration; qLabs®FIB Monitoring system; Clauss fibrinogen assay
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients giving birth in the Cochin Port Royal and Necker Enfants Malades (APHP) maternity units and cared for severe postpartum haemorrhage defined as bleeding greater than 1000 ml within 24 hours of postpartum, regardless of the route of delivery (vaginal delivery and cesarean section).
  Interventions: Biological: Fibrinogen concentration by the qLabs®FIB Monitoring system

INTERVENTIONS:
Biological: Fibrinogen concentration by the qLabs®FIB Monitoring system — A drop of blood (~15 μL) is taken from the blood sample for the complete haemostasis assessment (prothrombin level, activated partial thromboplastin time, fibrinogen). This assessment is part of the usual management of severe postpartum haemorrhage. It is carried out urgently in the hospital's medical biology laboratory at the start of treatment (T1) and during or at the end of treatment of the haemorrhage (T2). This drop of blood will allow the measurement of the fibrinogen concentration by the qLabs®FIB Monitoring system for the study at these two times.

SUMMARY:
In France in 2021, 11.6% of deliveries were complicated by a postpartum haemorrhage (PPH), including 3.0% by severe PPH (the bleeding volume exceeds 1000 ml). Severe PPH is the 5th cause of maternal death (8.4% or 1.2 deaths per 100,000 live births). These deaths were considered preventable in 90% of cases. A plasma fibrinogen concentration below 2 g/L is considered as a critical threshold which constitutes a marker of severity of PPH and is significantly associated with the occurrence of severe PPH. Measuring the concentration of fibrinogen using a rapid test, simple to perform and interpret, available in the delivery room could optimize the management of severe PPH. The qLabs®FIB analyzer distributed by the Stago Biocare laboratory for the rapid determination of the fibrinogen concentration at the patient's bedside could meet this objective.

DETAILED DESCRIPTION:
In France in 2021, 11.6% of deliveries were complicated by postpartum hemorrhage (PPH), including 3.0% by severe PPH (the bleeding volume exceeds 1000 ml). Severe PPH is the 5th cause of maternal death (8.4% or 1.2 deaths per 100,000 live births). These deaths were considered preventable in 90% of cases. A plasma fibrinogen concentration below 2 g/L is considered as a critical threshold which constitutes a marker of severity of PPH and is significantly associated with the occurrence of severe PPH. Measuring the concentration of fibrinogen using a rapid test, simple to perform and interpret, available in the delivery room could optimize the management of severe PPH. The qLabs®FIB analyzer distributed by Stago Biocare laboratory for the rapid determination of the fibrinogen concentration at the patient's bedside could meet this objective.

The hypothesis of the study is a concordance between the measurement of fibrinogen by the qLabs®FIB Monitoring system and by the Clauss fibrinogen assay in laboratory to identify patients with a fibrinogen level < 2 g/L.

The prospects are to provide an easy-to-use delocalized biology tool for early diagnosis of a fibrinogen concentration < 2g predictive of an unfavorable evolution in the context of severe PPH.

ELIGIBILITY:
Inclusion Criteria:

Adult patients having been informed of the study and not having objected to their participation and treated for severe postpartum haemorrhage defined as bleeding greater than 1000 ml within 24 hours postpartum, whatever the route delivery (vaginal route and caesarean section).

Exclusion Criteria:

* Opposition to participation in the study
* Presence of a constitutional fibrinogen deficiency
* Patients under guardianship or curatorship

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients giving birth in the two type 3 maternity wards of the Paris Center University Hospital Group : Necker-Enfants Malades et Cochin Port Royal (APHP) and with severe postpartum hemorrhage.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Agreement between fibrinogen measurement by qLabs®FIB and by the Clauss method | Through study completion, an average of 1 year
  Calculation of the average bias and the 95% limits of agreement between the measurement of qLabs®FIB fibrinogen in the delivery room and Clauss fibrinogen at the medical biology laboratory using the Bland and Altman graphic method. A difference of 0.1 g between the two techniques will be considered acceptable to identify patients with a fibrinogen level < 2 g/L.

SECONDARY OUTCOMES:
Evaluation of the ease of use of qLabs®FIB by the anesthesia team | Through study completion, an average of 1 year
  Ease of use of the qLabs®FIB assessed by a numerical scale between 0-10 by the anesthesia team.
Evaluation of the time taken to obtain the fibrinogen concentration using the 2 methods | Through study completion, an average of 1 year
  Time to obtain the fibrinogen result with the qLabs®FIB and the Clauss method at the medical biology laboratory using the emergency circuit proposed by the laboratory.
Evaluation of measurement failure by qLabs®FIB | Through study completion, an average of 1 year
  Number of failed fibrinogen measurements with qLabs®FIB defined as the absence of results returned by the monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Hawa KEITA-MEYER, MD-PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Marc SAMAMA, MD-PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hôpital Cochin Maternité Port Royal, Paris
  - Hôpital Necker-Enfants Malades, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sentilhes L, Vayssiere C, Deneux-Tharaux C, Aya AG, Bayoumeu F, Bonnet MP, Djoudi R, Dolley P, Dreyfus M, Ducroux-Schouwey C, Dupont C, Francois A, Gallot D, Haumonte JB, Huissoud C, Kayem G, Keita H, Langer B, Mignon A, Morel O, Parant O, Pelage JP, Phan E, Rossignol M, Tessier V, Mercier FJ, Goffinet F. Postpartum hemorrhage: guidelines for clinical practice from the French College of Gynaecologists and Obstetricians (CNGOF): in collaboration with the French Society of Anesthesiology and Intensive Care (SFAR). Eur J Obstet Gynecol Reprod Biol. 2016 Mar;198:12-21. doi: 10.1016/j.ejogrb.2015.12.012. Epub 2015 Dec 21. PMID 26773243
- [Background] Blondel B et al. Enquête nationale périnatale 2021
- [Background] Saucedo M, Tessier V, Leroux S, Almeras A, Deneux-Tharaux C. Mortalité maternelle en France, mieux comprendre pour mieux prévenir. Sages-Femmes. sept 2021;20(5):36-42
- [Background] Deneux-Tharaux C, Bouvier-Colle MH. Severe acute maternal morbidity in France: the epimoms population-based study. Am J Obstet Gynecol. 1 janv 2017;216(1):S345-6
- [Background] Godeberge C, Deneux-Tharaux C, Seco A, Rossignol M, Chantry AA, Bonnet MP; EPIMOMS Study Group. Maternal Intensive Care Unit Admission as an Indicator of Severe Acute Maternal Morbidity: A Population-Based Study. Anesth Analg. 2022 Mar 1;134(3):581-591. doi: 10.1213/ANE.0000000000005578. PMID 33989204
- [Background] Charbit B, Mandelbrot L, Samain E, Baron G, Haddaoui B, Keita H, Sibony O, Mahieu-Caputo D, Hurtaud-Roux MF, Huisse MG, Denninger MH, de Prost D; PPH Study Group. The decrease of fibrinogen is an early predictor of the severity of postpartum hemorrhage. J Thromb Haemost. 2007 Feb;5(2):266-73. doi: 10.1111/j.1538-7836.2007.02297.x. Epub 2006 Nov 6. PMID 17087729
- [Background] Deleu F, Deneux-Tharaux C, Chiesa-Dubruille C, Seco A, Bonnet MP; EPIMOMS study Group. Fibrinogen concentrate and maternal outcomes in severe postpartum hemorrhage: A population-based cohort study with a propensity score-matched analysis. J Clin Anesth. 2022 Oct;81:110874. doi: 10.1016/j.jclinane.2022.110874. Epub 2022 Jun 2. PMID 35662057
- [Background] Green L, Knight M, Seeney F, Hopkinson C, Collins PW, Collis RE, Simpson NA, Weeks A, Stanworth SJ. The haematological features and transfusion management of women who required massive transfusion for major obstetric haemorrhage in the UK: a population based study. Br J Haematol. 2016 Feb;172(4):616-24. doi: 10.1111/bjh.13864. Epub 2015 Dec 18. PMID 26683982
- [Background] Cortet M, Deneux-Tharaux C, Dupont C, Colin C, Rudigoz RC, Bouvier-Colle MH, Huissoud C. Association between fibrinogen level and severity of postpartum haemorrhage: secondary analysis of a prospective trial. Br J Anaesth. 2012 Jun;108(6):984-9. doi: 10.1093/bja/aes096. Epub 2012 Apr 6. PMID 22490316
- [Background] Ducloy-Bouthors AS, Mercier FJ, Grouin JM, Bayoumeu F, Corouge J, Le Gouez A, Rackelboom T, Broisin F, Vial F, Luzi A, Capronnier O, Huissoud C, Mignon A; FIDEL working group. Early and systematic administration of fibrinogen concentrate in postpartum haemorrhage following vaginal delivery: the FIDEL randomised controlled trial. BJOG. 2021 Oct;128(11):1814-1823. doi: 10.1111/1471-0528.16699. Epub 2021 Apr 7. PMID 33713384
- [Background] Liew-Spilger AE, Sorg NR, Brenner TJ, Langford JH, Berquist M, Mark NM, Moore SH, Mark J, Baumgartner S, Abernathy MP. Viscoelastic Hemostatic Assays for Postpartum Hemorrhage. J Clin Med. 2021 Aug 31;10(17):3946. doi: 10.3390/jcm10173946. PMID 34501395
- [Background] Huissoud C, Carrabin N, Audibert F, Levrat A, Massignon D, Berland M, Rudigoz RC. Bedside assessment of fibrinogen level in postpartum haemorrhage by thrombelastometry. BJOG. 2009 Jul;116(8):1097-102. doi: 10.1111/j.1471-0528.2009.02187.x. Epub 2009 May 12. PMID 19459866
- [Background] Collins PW, Cannings-John R, Bruynseels D, Mallaiah S, Dick J, Elton C, Weeks AD, Sanders J, Aawar N, Townson J, Hood K, Hall JE, Collis RE. Viscoelastometric-guided early fibrinogen concentrate replacement during postpartum haemorrhage: OBS2, a double-blind randomized controlled trial. Br J Anaesth. 2017 Sep 1;119(3):411-421. doi: 10.1093/bja/aex181. PMID 28969312
- [Background] Jokinen S, Kuitunen A, Uotila J, Yli-Hankala A. Thromboelastometry-guided treatment algorithm in postpartum haemorrhage: a randomised, controlled pilot trial. Br J Anaesth. 2023 Feb;130(2):165-174. doi: 10.1016/j.bja.2022.10.031. Epub 2022 Dec 7. PMID 36496259
- [Background] Sanfilippo S, Buisson L, Rouabehi H, Dujaric ME, Donnet T, de Raucourt E, Dumont B, Peynaud-Debayle E. The qLabs(R) FIB system, a novel point-of-care technology for a rapid and accurate quantification of functional fibrinogen concentration from a single drop of citrated whole blood. Thromb Res. 2023 Jun;226:159-164. doi: 10.1016/j.thromres.2023.03.018. Epub 2023 Apr 5. PMID 37178638